CLINICAL TRIAL: NCT06800833
Title: Effects of Mango or Low-Fat Cookie Consumption on Gut Health, and Its Relationship With Mental, Sexual and Skin Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB-25-0010
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gut Microbiome
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fat cookies (Active Comparator): Subjects consume 100 kcal of low-fat cookies daily for 4 weeks.
  Interventions: Other: Low fat cookies
- Mango (Experimental): Subjects consume 100 kcal of mango daily for 4 weeks.
  Interventions: Other: Mango

INTERVENTIONS:
Other: Low fat cookies — To determine the effects of low fat cookie consumption on physiological indicators of sexual, mental, skin, and gut health
  Arms: Low fat cookies
Other: Mango — To determine the effects of mango consumption on physiological indicators of sexual, mental, skin, and gut health
  Arms: Mango

SUMMARY:
The objective of the proposed research is to determine the effects of fresh mango consumption on gut microbiome, and its relationship with skin health, sexual and mental health in relatively healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects
* BMI 20-40 kg/m2

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required antibiotics use
* Required dietary supplement use
* Required medication of metabolic disorders, mental health and sexual health
* Allergy to mango or wheat

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of sexual health questionnaire scores | Baseline and week 4
  Change of sexual health questionnaire scores will be determined to examine effects of mango consumption vs low-fat cookies.
Change of depression questionnaire scores | Baseline and week 4
  Change of depression questionnaire scores will be determined to examine effects of mango consumption vs low-fat cookies.
Change of skin hydration scores | Baseline, 1 min post application and week 4consumption
  Change of skin hydration scores will be determined to examine effects of mango consumption vs low-fat cookies
Change of microbiome diversity | Baseline and week 4
  Change of microbiome diversity will be determined to examine effects of mango consumption vs low-fat cookies.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided